CLINICAL TRIAL: NCT00806286
Title: Phase 2 Randomized Study of Carboplatin/Paclitaxel With or Without CS-7017 in Chemotherapy-Naïve Subjects With Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of Carboplatin/Paclitaxel With or Without Investigational Drug (CS-7017) in Subjects With Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS7017-A-U202
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — efatutazone; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CS-7017 with Paclitaxel and Carboplatin (Experimental)
  Interventions: Drug: CS7017 tablets; Drug: Paclitaxel; Drug: Carboplatin
- Paclitaxel and Carboplatin (Placebo Comparator)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Placebo Tablets

INTERVENTIONS:
Drug: CS7017 tablets — CS7017 tablets, strength 0.25 mg, two tablets, two times daily for twenty-five to thirty months
  Arms: CS-7017 with Paclitaxel and Carboplatin
Drug: Paclitaxel — Intravenous (IV), 200 mg/m^2, once every three weeks for up to 18 weeks
Drug: Carboplatin — IV, area under the curve (AUC) of 6, once every three weeks for up to 18 weeks
Drug: Placebo Tablets — Placebo tablets matching CS-7017 tablets
  Arms: Paclitaxel and Carboplatin

SUMMARY:
The study has a safety and a Phase 2 portion. In the safety portion of the study, subjects with metastatic non-small cell lung cancer will be treated with study drug (CS-7017) in combination with carboplatin and paclitaxel to evaluate safety. In the Phase 2 portion of the study, subjects will receive study drug (CS-7017) or placebo in combination with carboplatin and paclitaxel to evaluate effectiveness and safety. The study will find out if adding CS-7017 to carboplatin and paclitaxel will be safe and improve progression free survival in subjects with metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic (stage IV) NSCLC with no significant pleural effusion or pleural involvement from the tumor
* Age greater than or equal to 18 years
* Adequate organ and bone marrow function

Exclusion Criteria:

* Any prior systemic therapy for NSCLC
* Major surgical procedure or other investigational agents within 4 weeks before study enrollment
* Need for concomitant use of other thiazolidinediones during the study
* History of any of the following conditions within 6 months prior to initiating study treatment: Diabetes mellitus requiring treatment with insulin or sulfonylureas or thiazolidinediones (TZDs) agents; Myocardia infarction with significant impairment of cardia function; Malabsorption syndrome, chronic diarrhea, inflammatory bowel disease or partial bowel obstruction;
* Clinically active brain metastases, uncontrolled seizure disorder; spinal cord compression or carcinomatous meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-12; Primary Completion 2012-01 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (27):
- United States (10):
  - University Colorado Cancer Center, Aurora, Colorado
  - Georgetown Univ. Medical Center, Washington D.C., District of Columbia
  - Southern Illinois Hematology/Oncology, Centralia, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Michiana Hematology-Oncology, South Bend, Indiana
  - Harbor View Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Penn State Milton Hershey Cancer Center, Hershey, Pennsylvania
  - Eastern Virginia Medical School, Norfolk, Virginia
- India (9):
  - Kidwai Memorial Institute of Oncology, Bangalore, Karnataka
  - Pentagon Research, Aundh, Maharashtra
  - Shatabdi Super Specialty Hospital, Nashik, Mumbai Naka
  - Hemato-Oncology Clinic, Vedanta, Gujarat, Navrangpura, Ahmedabad
  - Meenakshi Mission Hospital, Madurai, Tamil Nadu
  - Orchid Nursing Home, Kolkata, West Bengal
  - Apollo Specialty Hospital, Chennai
  - Ruby Hall Clinic, Pune
  - Noble Hospital, Pune
- Poland (3):
  - Oddzial Chemioterapii ZOZ MSWiA, Olsztyn
  - Oddzial Onkologii Klinicznej z Pododdzialem Dziennej Chemioterapii, Poznan
  - Specjalistyczny Szpital im. Prof. Alfresa Sokolowskiego, Szczecin
- Romania (5):
  - Oncomed SRL, Timișoara, Judet Timis
  - Spitalul Municipal Ploiesti, Ploieşti, Prahova
  - Institutul Oncologic Prof. Dr. Alexandru Trestioreanu, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca
  - Centrul de Oncologie Medicala, Iași

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 108 participants who met all inclusion and no exclusion criteria were randomized to CS-7017 or placebo combined with carboplatin/paclitaxel in the Phase 2 portion study. Three participants were enrolled in the Safety portion and received CS-7017 combined with carboplatin/paclitaxel (cycles 1-6) or CS-7017 monotherapy (subsequent cycles).
Groups:
- CS7017+Carboplatin+Paclitaxel: Participants who received CS-7017 by mouth (PO) approximately every 12 hours combined with carboplatin and paclitaxel administered IV once every 3 weeks (Day 1 each cycle).
- CS7017-matching Placebo+Carboplatin+Paclitaxel: Participants who received CS-7017-matching placebo by mouth (PO) approximately every 12 hours combined with carboplatin and paclitaxel administered IV once every 3 weeks (Day 1 each cycle).
- Safety Portion: Participants who received CS-7017 combined with carboplatin/paclitaxel (cycles 1-6) or CS-7017 monotherapy (subsequent cycles).
Period: Overall Study
Arm/Group | CS7017+Carboplatin+Paclitaxel | CS7017-matching Placebo+Carboplatin+Paclitaxel | Safety Portion
Started | 54 | 54 | 3
Completed | 0 | 0 | 0
Not Completed | 54 | 54 | 3
Not completed — Adverse Event | 5 | 2 | 0
Not completed — Disease progression | 31 | 38 | 1
Not completed — Death | 1 | 6 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 8 | 3 | 1
Not completed — Physician Decision | 2 | 2 | 0
Not completed — Due to a variety of reasons | 7 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CS7017+Carboplatin+Paclitaxel | CS7017-matching Placebo+Carboplatin+Paclitaxel | Safety Portion | Total
Number analyzed (Participants) | 54 | 54 | 3 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 48 | 39 | 1 | 88
  >=65 years | 6 | 15 | 2 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (8.19) | 59.4 (10.60) | 65.3 (12.01) | 58.4 (9.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 1 | 31
  Male | 41 | 37 | 2 | 80
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 22 | 22 | 0 | 44
  United States | 12 | 12 | 3 | 27
  Poland | 7 | 6 | 0 | 13
  India | 13 | 14 | 0 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-Free Survival at 18 Weeks Following Administration of Carboplatin/Paclitaxel With or Without CS-7017 in Chemotherapy-naïve Participants With Metastatic Non-small Cell Lung Cancer
Description: Progression-free survival (PFS) was defined as the time from the date of randomization to the earlier of the dates of the first objective documentation of disease progression (based upon radiographic tumor assessments) or death. As per Response Evaluation Criteria for Solid Tumors v1.0, disease progression was characterized as confirmed complete response (CR) defined as disappearance of all target lesions, confirmed partial response (PR) defined as ≥30% decrease from baseline, stable disease (SD) defined as neither progressive disease (PD) nor PR, and PD defined as ≥20% increase from smallest sum of longest diameter recorded since treatment started.
Time Frame: 18 weeks postdose
Population: Progression-free survival rates were assessed in the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CS7017+Carboplatin+Paclitaxel | CS7017-matching Placebo+Carboplatin+Paclitaxel
Number analyzed (Participants) | 54 | 54
percentage of participants | 40.2 [25.7 to 54.2] | 63.3 [48.7 to 74.9]
Statistical Analysis 1: Comparison: CS7017+Carboplatin+Paclitaxel vs CS7017-matching Placebo+Carboplatin+Paclitaxel; Test type: Superiority; p < 0.0001, Z-test — Two-sided p-value is calculated by dividing the square of the treatment group difference on the log-log scale by the standard error of the difference and referring the result to the standard normal distribution; Mean Difference (Final Values) = -23.2 — The estimated value represents the difference in treatments (%)
Statistical Analysis 2: Comparison: CS7017+Carboplatin+Paclitaxel vs CS7017-matching Placebo+Carboplatin+Paclitaxel; Test type: Superiority; p = 0.0499, Regression, Cox; Cox Proportional Hazard = 1.579, 95% CI 2-sided [1.0 to 2.5]

2. Primary Outcome: Percentage of Participants With Progression-Free Survival Based on Radiologic and Clinical Assessments and Death After Carboplatin/Paclitaxel With or Without CS-7017 in Chemotherapy-naïve Participants With Metastatic Non-small Cell Lung Cancer
Description: Progression-free survival (PFS) was defined as the time from the date of randomization to the earlier of the dates of the first objective documentation of disease progression (based upon radiographic tumor assessments) or death. Disease progression was determined in accordance with the RECIST version 1.0 criteria.
Time Frame: 18 weeks postdose
Population: Progression-free survival rates were assessed in the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CS7017+Carboplatin+Paclitaxel | CS7017-matching Placebo+Carboplatin+Paclitaxel
Number analyzed (Participants) | 54 | 54
percentage of participants | 37.9 [23.5 to 52.1] | 63.3 [48.7 to 74.9]
Statistical Analysis 1: Comparison: CS7017+Carboplatin+Paclitaxel vs CS7017-matching Placebo+Carboplatin+Paclitaxel; Test type: Superiority — Two-sided p-value is calculated by dividing the square of the treatment group difference on the log-log scale by the standard error of the difference and referring the result to the standard normal distribution; p < 0.0001, Z-test; Mean Difference (Final Values) = -25.5 — The estimated value represents the difference in treatments (%)

3. Secondary Outcome: Summary of Kaplan-Meier Analysis of Overall Survival Following Administration of Carboplatin/Paclitaxel With or Without CS-7017 in Chemotherapy-naïve Participants With Metastatic Non-small Cell Lung Cancer
Description: Overall survival (OS) is defined as the time from randomization to the date of death resulting from any cause.
Time Frame: Baseline to date of death, up to approximately 2 years postdose
Population: OS was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CS7017+Carboplatin+Paclitaxel | CS7017-matching Placebo+Carboplatin+Paclitaxel
Number analyzed (Participants) | 54 | 54
days | 244.0 [158.0 to 353.0] | 292.0 [233.0 to 404.0]

4. Secondary Outcome: Number of Participants With Best Overall Tumor Response and Objective Response Rate Following Administration of Carboplatin/Paclitaxel With or Without CS-7017 in Chemotherapy-naïve Participants With Metastatic Non-small Cell Lung Cancer
Description: As per Response Evaluation Criteria for Solid Tumors v1.0, the best overall response was characterized as confirmed complete response (CR) defined as disappearance of all target lesions, confirmed partial response (PR) defined as ≥30% decrease from baseline, stable disease (SD) defined as neither progressive disease (PD) nor PR, and PD defined as ≥20% increase from smallest sum of longest diameter recorded since treatment started. Objective response rate (ORR) was defined as CR + PR.
Time Frame: Baseline to disease progression, death, or withdrawal from study, up to approximately 2 years postdose
Population: Best overall response was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS7017+Carboplatin+Paclitaxel | CS7017-matching Placebo+Carboplatin+Paclitaxel
Number analyzed (Participants) | 54 | 54
Participants
  Confirmed complete response (CR) | 0 | 0
  Confirmed partial response (PR) | 11 | 16
  Objective response (Confirmed CR+PR) | 11 | 16
  Stable disease (SD) | 11 | 18
  Progressive disease (PD) | 17 | 5
  Unknown | 8 | 7
  Best Objective Response of SD or Better | 29 | 42

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events Related to CS-7017/Placebo Following Administration of Carboplatin/Paclitaxel With or Without CS-7017 in Chemotherapy-naïve Participants With Metastatic Non-small Cell Lung Cancer
Time Frame: Baseline up to approximately 2 years postdose
Population: Treatment-emergent adverse events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CS7017+Carboplatin+Paclitaxel | CS7017-matching Placebo+Carboplatin+Paclitaxel | Safety Portion
Number analyzed (Participants) | 54 | 54 | 3
Participants
  Any TEAE | 42 | 25 | 3
  Blood and Lymphatic System Disorders | 10 | 11 | 3
  Anaemia | 7 | 5 | 2
  Febrile neutropenia | 2 | 0 | 0
  Leukopenia | 1 | 2 | 0
  Lymphopenia | 0 | 2 | 0
  Neutropenia | 2 | 3 | 2
  Pancytopenia | 1 | 0 | 0
  Thrombocytopenia | 5 | 4 | 1
  Cardiac Disorders | 2 | 0 | 0
  Acute myocardial infarction | 1 | 0 | 0
  Palpitations | 1 | 0 | 0
  Gastrointestinal Disorders | 10 | 7 | 2
  Abdominal pain | 1 | 1 | 0
  Abdominal pain upper | 0 | 1 | 0
  Constipation | 1 | 0 | 1
  Diarrhoea | 1 | 5 | 0
  Dry mouth | 1 | 1 | 0
  Dyspepsia | 1 | 0 | 0
  Gastrooesophageal reflux disease | 2 | 0 | 0
  Hypoaesthesia oral | 1 | 0 | 0
  Melaena | 1 | 0 | 0
  Mouth haemorrhage | 1 | 0 | 0
  Nausea | 5 | 3 | 2
  Pancreatitis | 0 | 1 | 0
  Stomatitis | 1 | 0 | 0
  Vomiting | 2 | 2 | 0
  General Disorders & Administration Site Conditions | 34 | 16 | 3
  Asthenia | 2 | 3 | 0
  Chest pain | 1 | 0 | 0
  Chills | 0 | 0 | 1
  Edema event | 31 | 12 | 3
  Fatigue or Asthenia event | 12 | 9 | 2
  Fatigue | 11 | 7 | 2
  Generalised oedema | 2 | 0 | 1
  Localised oedema | 1 | 0 | 0
  Malaise | 0 | 0 | 1
  Oedema | 5 | 1 | 0
  Oedema peripheral | 14 | 8 | 0
  Pyrexia | 1 | 1 | 0
  Immune System Disorders | 1 | 0 | 0
  Hypersensitivity | 1 | 0 | 0
  Infections and Infestations | 1 | 0 | 0
  Infection | 1 | 0 | 0
  Investigations | 16 | 7 | 2
  Alanine aminotransferase increased | 0 | 1 | 0
  Aspartate aminotransferase increased | 0 | 0 | 1
  Blood alkaline phosphatase increased | 0 | 2 | 0
  Blood creatinine increased | 2 | 0 | 0
  Transaminases increased | 0 | 1 | 0
  Weight decreased | 1 | 1 | 0
  Weight increased | 15 | 3 | 2
  Metabolism and Nutrition Disorders | 10 | 11 | 2
  Anorexia | 5 | 6 | 1
  Dehydration | 0 | 1 | 0
  Fluid retention | 2 | 1 | 0
  Hypercholesterolaemia | 4 | 1 | 1
  Hyperglycaemia | 0 | 1 | 0
  Hypermagnesaemia | 0 | 1 | 0
  Hypertriglyceridaemia | 3 | 1 | 0
  Hypocalcaemia | 0 | 1 | 0
  Hyponatraemia | 0 | 2 | 0
  Musculoskeletal and Connective Tissue Disorders | 1 | 0 | 1
  Bone pain | 1 | 0 | 0
  Joint swelling | 0 | 0 | 1
  Nervous System Disorders | 2 | 3 | 1
  Dizziness | 1 | 1 | 0
  Dysgeusia | 1 | 0 | 0
  Guillain-Barre Syndrome | 0 | 1 | 0
  Neuropathy peripheral | 0 | 0 | 1
  Paraesthesia | 0 | 1 | 0
  Renal and Urinary Disorders | 2 | 0 | 0
  Haematuria | 1 | 0 | 0
  Urinary retention | 1 | 0 | 0
  Respiratory, Thoracic, and Mediastinal Disorders | 12 | 2 | 0
  Cough | 2 | 0 | 0
  Dyspnoea | 4 | 0 | 0
  Haemoptysis | 1 | 0 | 0
  Pleural effusion | 5 | 0 | 0
  Pleurisy | 2 | 1 | 0
  Pulmonary congestion | 0 | 1 | 0
  Respiratory distress | 1 | 0 | 0
  Wheezing | 1 | 0 | 0
  Skin and Subcutaneous Tissue Disorders | 6 | 3 | 0
  Acne | 1 | 0 | 0
  Alopecia | 1 | 1 | 0
  Pruritus | 0 | 1 | 0
  Rash | 0 | 2 | 0
  Rash erythematous | 1 | 0 | 0
  Skin lesion | 1 | 0 | 0
  Swelling face | 3 | 0 | 0
  Vascular Disorders | 1 | 1 | 0
  Hypotension | 0 | 1 | 0
  Pallor | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from baseline to the end of study assessment, approximately 2 years post dose.
Description: An adverse event (AE) is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. All-cause mortality includes all deaths that occurred during the study and within 30 days after the last dose of study drug.
Arm/Group | CS7017+Carboplatin+Paclitaxel | CS7017-matching Placebo+Carboplatin+Paclitaxel | Safety Portion
All-Cause Mortality (participants affected / at risk) | 8/54 | 14/54 | 0/3
Serious Adverse Events (participants affected / at risk) | 27/54 | 29/54 | 1/3
Other Adverse Events (participants affected / at risk) | 53/54 | 53/54 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CS7017+Carboplatin+Paclitaxel (N=54) | CS7017-matching Placebo+Carboplatin+Paclitaxel (N=54) | Safety Portion (N=3)
Anaemia (Blood and lymphatic system disorders) | 5 | 6 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Death (General disorders) | 2 | 2 | 0
Disease progression (General disorders) | 4 | 7 | 0
Edema event (General disorders) | 1 | 0 | 0
Fatigue or Asthenia event (General disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bacteria stool identified (Investigations) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Guillain-Barre Syndrome (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CS7017+Carboplatin+Paclitaxel (N=54) | CS7017-matching Placebo+Carboplatin+Paclitaxel (N=54) | Safety Portion (N=3)
Anaemia (Blood and lymphatic system disorders) | 40 | 27 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 12 | 9 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 15 | 22 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 18 | 2
Tachycardia (Cardiac disorders) | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 0
Constipation (Gastrointestinal disorders) | 9 | 8 | 1
Diarrhoea (Gastrointestinal disorders) | 13 | 13 | 0
Nausea (Gastrointestinal disorders) | 18 | 8 | 2
Vomiting (Gastrointestinal disorders) | 8 | 12 | 0
Asthenia (General disorders) | 8 | 7 | 0
Chest pain (General disorders) | 9 | 10 | 0
Chills (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 4 | 7 | 0
Edema event (General disorders) | 32 | 13 | 3
Fatigue or Asthenia event (General disorders) | 24 | 20 | 3
Fatigue (General disorders) | 18 | 14 | 3
Generalised oedema (General disorders) | 2 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 5 | 2 | 0
Oedema peripheral (General disorders) | 15 | 9 | 0
Pain (General disorders) | 4 | 2 | 0
Pyrexia (General disorders) | 5 | 10 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 3 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 1
Protein total decreased (Investigations) | 0 | 0 | 1
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 6 | 0
Weight increased (Investigations) | 16 | 3 | 2
Anorexia (Metabolism and nutrition disorders) | 9 | 10 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 5 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No